CLINICAL TRIAL: NCT02582294
Title: Description of Obstetrical Care, Mainly Anesthesic, in Patients With Fabry's Disease
Brief Title: Fabry's Disease and Pregnancy (PREFAB)
Acronym: PREFAB
Status: Terminated | Type: Observational
Why Stopped: Difficulty in patient recruitment
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Sponsor
Other Study IDs: OLE_2015_4
Record Dates: First submitted 2015-10-15; First posted 2015-10-21 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Fabry's Disease; Pregnancy
MeSH Terms: conditions — Fabry Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Questionnaire

SUMMARY:
Fabry's disease is a progressive systemic disease X-linked which combines neurological (Fabry's pain crises), dermatologic (angiokeratomas), renal (renal failure), cardiovascular (hypertrophic cardiomyopathy, valvular disease, conduction disorder, coronary heart disease) and cerebral vascular (stroke) symptoms .

It is a glycosphingolipid metabolism disorder due to deficient or absent activity of the alpha-galactosidase A, causing accumulation of globotriaosylceramide in the lysosomes.

The incidence is estimated being 1/40 000. Some patients suffering from Fabry's disease today are of childbearing age and their multidisciplinary care (by neurologists, obstetricians and anesthetists) raises several questions.

About the anesthetic, the question of epidural block is debated in patients with neurological diseases and recommendations are not unequivocal.

Indeed one of the problems of the management in those conditions is the potential worsening of the disease because of the anesthetic procedure. In addition, the possibility of an antiplatelet and / or an anticoagulant treatment in these patients may also contre-indicate an epidural block.

The rate of epidural block achieved in patients with Fabry's disease is not currently known. Moreover, only sparse data on pregnancy outcomes in these patients are reported.

ELIGIBILITY:
Inclusion Criteria:

* Fabry's disease patients, aged 18 years or more, having had at least one childbirth

Exclusion Criteria:

* Patient under a legal protection procedure
* Patient denying to participate to the study
* Lack of affiliation to a social security system

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Fabry's disease patients having had at least one childbirth
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Proportion of Fabry's disease patients having had an epidural block in childbirth. | The duration of the interview for this study with women with Fabry disease's will be one hour

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe hospitalier Diaconesses Croix Saint Simon, Paris, Île-de-France Region, France